CLINICAL TRIAL: NCT01873963
Title: Genotype-Phenotype Associations in Pediatric Cardiomyopathy
Brief Title: Genotype-Phenotype Associations in Pediatric Cardiomyopathy (PCM GENES)
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: Carelon Research (Other); Children's Hospital Medical Center, Cincinnati (Other); Washington University School of Medicine (Other); Children's Hospital of Philadelphia (Other); Columbia University (Other); Boston Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Primary Children's Hospital (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); Stollery Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Miami (Other); Children's Hospital Colorado (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Steve Lipshultz, Schotanus Family Endowed Chair of Pediatrics, Professor and Chair, Carman and Ann Adams Department of Pediatrics, Wayne State University School of Medicine; President, University Pediatricians and Pediatrician-in-Chief, Children's Hospital of Michigan, Wayne State University
Other Study IDs: 1R01HL111459-01 (NIH); 1R01HL111459-01 (NIH)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Restrictive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio specimen blood samples were collected for patients enrolled in the PCM Genes study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric cardiomyopathy: Diagnosis of primary or idiopathic dilated, hypertrophic or restrictive cardiomyopathy. Diagnosis must have been made before the age of 18 and must be confirmed by established echocardiographic criteria or cardiac MRI (cMRI) at the time of diagnosis.

SUMMARY:
Cardiomyopathy in children is a serious disease which can result in death, disability, heart transplantation or serious heart rhythm disorders. Doctors know little about the causes of cardiomyopathy but would like to learn more. In fact, up to 50-75% of cases in children have no known cause. For this reason, the purpose of this study is to identify genes that cause cardiomyopathy or that influence how people with cardiomyopathy do over time. These findings could improve disease prevention, surveillance, early management, and prognosis.

DETAILED DESCRIPTION:
Pediatric cardiomyopathy is a heterogeneous genetic disease with high morbidity and mortality in which children often present with fulminant disease leading to death or transplant. The long-term goal of this project is to identify the genetic basis of cardiomyopathy and to correlate these findings with clinical phenotypes for risk stratification. These findings could improve disease prevention, surveillance, early management, and prognosis.

The specific aims of this study are:

1. To identify the disease-causing and disease-associated genetic variants underlying pediatric cardiomyopathy in a carefully phenotyped cohort.
2. To identify genotype-phenotype correlations that allow for risk stratification and improve management and therapy.

Exome sequencing will be used as part of a tiered genetic analysis in a large cohort of up to 700 pediatric cardiomyopathy subjects with systolic (dilated cardiomyopathy) or diastolic (hypertrophic or restrictive cardiomyopathy) dysfunction. The biological parent(s) of enrolled participants will also be approached about participating and providing a blood sample for genetic testing. In addition to the parent(s), the participants siblings and other relatives may also be approached regarding enrollment, based on the pedigree and family history.

This study will significantly increase our understanding of pediatric cardiomyopathy by defining the prevalence of mutations in genes known to cause cardiomyopathy as well as identifying novel disease-causing genes in the pediatric population. Genetic association tests will identify variants that modify disease. Novel bioinformatics and systems biology applications for interpretation of exome level genetic information will contribute fundamental knowledge and technical innovation to the translation of genomic data to clinical utility. These aims will provide critical genetic architecture data, identify variants with large effects, and enable genotype-phenotype correlations necessary for advancing management and therapy.

The Study will have two components: 1) clinical data collection by chart review and family interview, and 2) biospecimen collection and genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient is alive. (except samples from deceased relatives who have consented for testing).Patients who are status-post heart transplant are eligible if pre-transplant longitudinal data are available.
* Under age 18 years at the time of diagnosis of either primary or idiopathic dilated, hypertropic, or restrictive cardiomyopathy.
* A diagnosis of cardiomyopathy which, at the time of diagnosis, was confirmed by echocardiographic criteria or cardiac MRI

Exclusion Criteria:

A patient is not eligible for enrollment if one or more of the following conditions are met at the time of presentation with cardiomyopathy:

* Arrhythmogenic right ventricular dysplasia
* Neuromuscular disease (defined by specific conditions)
* Endocrine disease known to cause heart muscle disease (including infants of diabetic mothers)
* History of rheumatic fever
* Toxic exposures known to cause heart muscle disease (anthracyclines, mediastinal radiation, iron overload or heavy metal exposure)
* HIV infection or born to an HIV positive mother
* Kawasaki disease
* Immunologic disease
* Invasive cardiothoracic procedures or major surgery during the preceding month, except those specifically related to cardiomyopathy including left ventricular assist device (LVAD), extracorporeal membrane oxygenator (ECMO), and automatic implantable cardioverter/defibrillator (AICD) placement.
* Uremia, active or chronic
* Abnormal ventricular size or function that can be attributed to intense physical training or chronic anemia
* Chronic arrhythmia, unless there are studies documenting inclusion criteria prior to the onset of arrhythmia (except a patient with chronic arrhythmia, subsequently ablated, whose cardiomyopathy persists after two months is not to be excluded).
* Malignancy
* Systemic Hypertension
* Pulmonary parenchymal or vascular disease (e.g., cystic fibrosis, cor pulmonale, or pulmonary hypertension)
* Ischemic coronary vascular disease
* Association with drugs known to cause hypertrophy (e.g., growth hormone, corticosteroids, cocaine)
* Genetic syndrome or chromosomal abnormality known to be associated with cardiomyopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric cases of dilated, hypertrophic or restrictive cardiomyopathy and select relatives will be enrolled at 11 pediatric cardiology centers in the US and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2013-04; Primary Completion 2017-02 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Time to death | 2 years

SECONDARY OUTCOMES:
Time to transplant | 2 years
Time to normalized left ventricular size or function in dilated cardiomyopathy | 2 years
Septal:Posterior wall thickness ratio in hypertrophic cardiomyopathy | 2 years
Left ventricular outflow tract in hypertrophic cardiomyopathy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Lipshultz, MD, Principal Investigator — Wayne State University
Locations (12):
- United States (11):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital of New York, Columbia Presbyterian Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Primary Children's Medical Center, Salt Lake City, Utah
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ware SM, Wilkinson JD, Tariq M, Schubert JA, Sridhar A, Colan SD, Shi L, Canter CE, Hsu DT, Webber SA, Dodd DA, Everitt MD, Kantor PF, Addonizio LJ, Jefferies JL, Rossano JW, Pahl E, Rusconi P, Chung WK, Lee T, Towbin JA, Lal AK, Bhatnagar S, Aronow B, Dexheimer PJ, Martin LJ, Miller EM, Sleeper LA, Razoky H, Czachor J, Lipshultz SE; Pediatric Cardiomyopathy Registry Study Group. Genetic Causes of Cardiomyopathy in Children: First Results From the Pediatric Cardiomyopathy Genes Study. J Am Heart Assoc. 2021 May 4;10(9):e017731. doi: 10.1161/JAHA.120.017731. Epub 2021 Apr 28. PMID 33906374